CLINICAL TRIAL: NCT04541355
Title: A Phase II Study of Sodium Thiosulfate (STS) for Prevention of Ototoxicity in Patients With Locally Advanced Squamous Cell Carcinoma of Head and Neck (SCCHN) Undergoing Concurrent Chemoradiation With Cisplatin
Brief Title: Sodium Thiosulfate in Preventing Ototoxicity for Squamous Cell Cancer Patients Undergoing Chemoradiation With Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hyunseok Kang, MD (Other)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor-Investigator, Hyunseok Kang, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20208; NCI-2020-05752 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Clinical Stage III Human Papillomavirus (HPV)-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Locally Advanced Head and Neck Squamous Cell Carcinoma; Locally Advanced Hypopharyngeal Squamous Cell Carcinoma; Locally Advanced Laryngeal Squamous Cell Carcinoma; Locally Advanced Oral Cavity Squamous Cell Carcinoma; Locally Advanced Oropharyngeal Squamous Cell Carcinoma; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Lip and Oral Cavity Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVC Hypopharyngeal Carcinoma AJCC v8; Stage IVC Laryngeal Cancer AJCC v8; Stage IVC Lip and Oral Cavity Cancer AJCC v8; Stage IVC Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Radiotherapy; Radiation; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin, Radiotherapy, STS (Experimental): Patients undergo standard of care radiation therapy daily in combination with cisplatin on day 1. Between 4-5 hours after each cisplatin infusion, patients also receive sodium thiosulfate over 1-2 hours on day 1. Treatment will continue on either a 1 week or 3 week cycle per physician discretion for up to 6-7 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Other: Hearing Handicap Inventory for Adults - Screening; Radiation: Radiation Therapy; Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; Lederplatin; Metaplatin; Neoplatin; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platiran; Platistin; Platosin
Other: Hearing Handicap Inventory for Adults - Screening — Patient self-assessment questionnaire to measure probability of hearing impairment
Radiation: Radiation Therapy — Radiation therapy will be delivered according to the standard of care
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, Not otherwise specified (NOS); Radiotherapeutics; Radiotherapy; RT
Drug: Sodium Thiosulfate — Given IV
  Other Names: Cyanide Antidote Package; Disodium Thiosulfate; S-Hydril; Sodium Hyposulfate; Sodium Thiosulfate Pentahydrate; Sodium Thiosulphate; Sodothiol; Thiosulfate, Sodium, Pentahydrate; Thiosulfuric Acid Disodium Salt

SUMMARY:
This phase II trial investigates how well sodium thiosulfate works in preventing ototoxicity (hearing loss/damage) in patients with squamous cell cancer of the head and neck that has spread to nearby tissue or lymph nodes (locally advanced) who are undergoing a chemoradiation. Sodium thiosulfate is a type of medication used to treat cyanide poisoning and to help lessen the side effects from cisplatin. Chemotherapy drugs, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy with radiation therapy may kill more tumor cells. The purpose of this trial is to find out whether it is feasible to give sodium thiosulfate 4 hours after each cisplatin infusion along with standard of care radiation therapy in patients with head and neck cancer. Giving sodium thiosulfate after cisplatin may help decrease the risk of hearing loss.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish feasibility of intravenous sodium thiosulfate (STS) after each dose of concurrent cisplatin in patients with locally advanced head and neck squamous cell carcinoma undergoing definitive radiotherapy.

SECONDARY OBJECTIVES:

I. To determine the rate of grade >= 2 hearing impairment based on Common Terminology Criteria for Adverse Events (CTCAE) version 5 with use of STS after concurrent chemoradiation with cisplatin 3 months post-treatment.

II. To determine the rate of tinnitus measured by Patient Reported Outcomes (PRO)-CTCAE with use of STS 3 months post-treatment.

III. To describe patient reported outcomes with STS measured with PRO-CTCAE for selected oral, gastrointestinal (GI), neurologic and perceptual symptoms.

IV. To describe patient reported outcomes measured with Hearing Handicap Inventory for Adults - Screening (HHIA-S) compared to results from standard NRG Oncology head and neck trials (such as Radiation Therapy Oncology Group (RTOG) 1016).

OUTLINE:

Patients undergo standard of care radiation therapy in combination with cisplatin therapy for up to 6-7 weeks. Cisplatin treatment repeats weekly for up to 7 cycles, or every 21 days for up to 3 cycles. After each cisplatin infusion, patients also receive an infusion of sodium thiosulfate. The dosing schedule for cisplatin will be at the discretion of the treating physician.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed locoregionally advanced squamous cell carcinomas of mucosal surfaces of head and neck who are being treated with concurrent chemoradiation with cisplatin
2. Participants must be eligible for cisplatin-based concurrent chemotherapy in conjunction with at least 6 weeks of daily fractionated radiation therapy
3. Age >=18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
5. Demonstrates adequate organ function as defined below:

   1. Absolute neutrophil count >= 1,000/microliter (mcL)
   2. Platelets >= 100,000/mcL
   3. Total bilirubin within normal institutional limits, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits
   4. Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase (SGOT)) =< 3 X institutional upper limit of normal
   5. Alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase (SGPT)) =< 3 X institutional upper limit of normal
   6. Creatinine =< 1.5 x within institutional upper limit of normal OR creatinine clearance glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2, calculated using the Cockcroft-Gault equation, unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
6. Ability to understand a written informed consent document, and the willingness to sign it
7. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
8. The effects of sodium thiosulfate (STS) on the developing human fetus are unknown. For this reason and because cisplatin used in this trial are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception such as hormonal and/or barrier method of birth control for the duration of study participation and for 3 months after last administration of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after last administration of study treatment

Exclusion Criteria:

1. Participants that are not eligible for cisplatin-based chemoradiation for reasons such as chronic kidney disease, severe hearing loss, and severe peripheral neuropathy
2. Uncontrolled inter-current illness or psychiatric illness/social situation that would limit compliance with study requirements
3. Has known hypersensitivity to cisplatin, sodium thiosulfate or any of its excipients
4. Has profound hearing impairment at baseline and cannot hear a sound below 90 decibels (dB)
5. Participants with uncompensated congestive heart failure New York Heart Association (NYHA) class 3 or above
6. Participants who cannot get secure venous access using either a Mediport or a peripherally inserted central catheter (PICC) line for safe administration of intravenous sodium thiosulfate
7. Pregnant women are excluded from this study because cisplatin is a cytotoxic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cisplatin or sodium thiosulfate, breastfeeding should be discontinued if the mother is treated with either agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyunseok Kang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin, Radiotherapy, STS: Participants undergo standard of care radiation therapy daily in combination with cisplatin on day 1. Between 4-5 hours after each cisplatin infusion, patients also receive sodium thiosulfate over 1-2 hours on day 1. Treatment will continue on either a 1 week or 3 week cycle per physician discretion for up to 6-7 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cisplatin, Radiotherapy, STS
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin, Radiotherapy, STS
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 3
  50-59 years old | 6
  60-69 years old | 4
  70-79 years old | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Successfully Completed Planned Treatment
Description: Evaluated as the successful completion of at least 5 weekly cisplatin or 2 high dose cisplatin without any extended treatment related delays more than 7 days. Overall successful completion is defined as completion by at least 75% of patients.
Time Frame: Up to 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin, Radiotherapy, STS
Number analyzed (Participants) | 16
Participants | 15

2. Secondary Outcome: Proportion of Participants With Reported High Grade Ototoxicity
Description: The proportion of participants with a reported change of grade >= 2 hearing impairments based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (for patients on a monitoring program with audiogram) will be reported.
Time Frame: Up to 18 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Cisplatin, Radiotherapy, STS
Number analyzed (Participants) | 16
proportion of participants | 0.18

3. Secondary Outcome: Number of Participants Reporting Tinnitus by Severity
Description: The frequency of tinnitus will be measured by participants' worst level response at any time point on the PRO-CTCAE® question "In the last 7 days, what was the severity of ringing in your ears at its worst?". Item responses were categorized as 'None', 'Mild', 'Moderate', 'Severe', and 'Very Severe'.
Time Frame: Up to 18 weeks
Measure: Number; unit: participants
Arm/Group | Cisplatin, Radiotherapy, STS
Number analyzed (Participants) | 16
participants
  None | 4
  Mild | 7
  Moderate | 4
  Severe | 1
  Very Severe | 0

4. Secondary Outcome: Percentage of Participants Reporting Sodium Thiosulfate (STS)-Specific Symptomology
Description: The percentage of participants reporting STS specific adverse events will be measured by affirmative responses on the PRO-CTCAE® on any of the selected oral, gastrointestinal, neurologic and visual/perceptual symptoms.
Time Frame: Up to 18 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Cisplatin, Radiotherapy, STS
Number analyzed (Participants) | 16
percentage of participants | 100

5. Secondary Outcome: Frequency of Hearing Handicap
Description: The Hearing Handicap Inventory for Adults -Screener (HHIA-S), is a 10-item, self-assessment screening assessment developed to quickly determine the suggested level of hearing handicap. The participants respond to each of the items with a Yes (score of 4), Sometimes (score of 2), or No (score of 0). Total Scores are then summed for overall score (range 0-40) and then assigned a category for a suggested hearing handicap; 0-8 suggesting no handicap, 10-24 suggesting a mild-moderate handicap, and 26-40 suggesting significant hearing handicap. The frequency of participants for worse reported score will be reported
Time Frame: Up to 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin, Radiotherapy, STS
Number analyzed (Participants) | 16
Participants
  Suggesting no handicap | 11
  Suggesting a mild-moderate handicap | 5
  Suggesting significant hearing handicap | 0

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Arm/Group | Cisplatin, Radiotherapy, STS
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin, Radiotherapy, STS (N=16)
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin, Radiotherapy, STS (N=16)
Abdominal Pain (Gastrointestinal disorders) | 1
Allergic Reaction (Immune system disorders) | 1 — Hives
Anemia (Blood and lymphatic system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Aphonia (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Blood and lymphatic system disorders, Other (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Creatinine increased (Investigations) | 3
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 5
Dysgeusia (Nervous system disorders) | 7
Dysphagia (Gastrointestinal disorders) | 6
Ear Pain (Ear and labyrinth disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 3
Gastrointestinal disorders, Other (Gastrointestinal disorders) | 5
Headaches (Nervous system disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3
Investigations, Other (Investigations) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 4
Lymph Node Pain (Blood and lymphatic system disorders) | 2
Lymphocyte count decreased (Investigations) | 1
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Musculoskeletal, Other (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Neutrophil Count Decreased (Investigations) | 2
Oral pain (Gastrointestinal disorders) | 1
Paresthesia (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 6
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5
Trismus (Musculoskeletal and connective tissue disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight Loss (Metabolism and nutrition disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04541355/Prot_SAP_000.pdf